CLINICAL TRIAL: NCT03588481
Title: Evaluation of Effectiveness and Safety of DESyne X2 in Routine Clinical Practice; A Multicenter, Prospective Observational Study
Brief Title: IRIS- DESyne X2 in the IRIS-DES Registry
Acronym: IRIS DESyne X2
Status: Recruiting | Type: Observational
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, Professor, Division of Cardiology, Department of Medicine, Heart Institute, Asan Medical Center, University of Ulsan College of Medicine, Asan Medical Center
Organization: Asan Medical Center (Other)
Other Study IDs: AMCCV2018-09
Record Dates: First submitted 2018-07-05; First posted 2018-07-17 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Coronary Stenosis; Coronary Occlusion; Coronary Disease
Keywords: PCI; DES; real world
MeSH Terms: conditions — Coronary Stenosis; Coronary Occlusion; Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Coronary stenosis
  Interventions: Device: DESyne X2

INTERVENTIONS:
Device: DESyne X2 — Novolimus-eluting stent

SUMMARY:
This study evaluates effectiveness and safety of DESyne X2 in Routine Clinical Practice.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 and more
* Intervention with DeSyne X2 drug-eluting coronary stent
* Agreed with written informed consent form

Exclusion Criteria:

* Intervention with DeSyne X2 drug-eluting coronary stent and other drug eluting stent at the same time
* Life expectancy of 1year and under
* Cardiac shock

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with DeSyne X2 stent
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-11-28 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite event rate | 1year
  Death, non-fatal myocardial infarction, Target Vessel Revascularization

SECONDARY OUTCOMES:
All death | 5years
Cardiac death | 5years
Myocardial infarction | 5years
Composite event of death or myocardial infarction | 5years
Composite event of cardiac death or myocardial infarction | 5years
Target Vessel revascularization | 5years
Target Lesion revascularization | 5years
Stent thrombosis | 5years
  stent thrombosis as classified by an Academic Research Consortium
Stroke | 5years
Procedural success | 3days
  defined as achievement of a final diameter stenosis of <30% by visual estimation, without the occurrence of death, Q-wave MI, or urgent revascularization during the index hospitalization.

CONTACTS AND LOCATIONS:
Locations (6):
- South Korea (6):
  - Hallym Hospital, Incheon
  - Asan Medical Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - The Catholic University of Korea Seoul St. Mary's Hospital, Seoul
  - The Catholic University of Korea, Eunpyeong St. Mary's Hospital, Seoul
  - St.carollo Hospital, Suncheon

IPD SHARING:
Plan to Share IPD: Undecided